CLINICAL TRIAL: NCT05647031
Title: Pain in Competitive Athletes With Physical Disabilities and Techniques for Its Management
Status: Completed | Type: Observational
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Sandra Constantino Murillo, Principal Investigator, Universidad Politecnica de Madrid
Other Study IDs: UPMadrid
Record Dates: First submitted 2022-11-21; First posted 2022-12-12 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Athletic Injuries; Physical Disability; Chronic Pain
Keywords: Athlete; Physical disability; Competition; Chronic pain; Psychological models
MeSH Terms: conditions — Athletic Injuries; Chronic Pain | interventions — Methods

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 20 participants were interviewed on a voluntary basis: A total of 20 participants were interviewed on a voluntary basis (7 competitive athletes with 17 physical disabilities, 4 physiotherapists, 5 coaches and 4 psychologists)
  Interventions: Other: Qualitative study. Pain in competitive athletes with physical disabilities and techniques for its management.

INTERVENTIONS:
Other: Qualitative study. Pain in competitive athletes with physical disabilities and techniques for its management. — This study used a qualitative, exploratory and descriptive methodology, with a semi-structured interview technique. The purpose was to respond to the specific objectives set out in this research from the perspective of competitive athletes and sports agents (physiotherapist, coach and psychologist). The thematic cores that served as a script for the interview were for the athletes and sports agents 1) sporting characteristics of the professionals; 2) perception of how pain affects this type of athlete and what repercussions it has on the development of their sporting career, and 3) knowledge of techniques and/or strategies for pain management (athlete, coach and psychologist).
  The interviews were conducted via skype. After transcription of all the interviews, validation by the interviewees was applied for the reliability of the research. Two types of triangulation were applied to ensure the quality of the data.

SUMMARY:
There are psychosocial factors that affect pain, and therefore, psychological intervention techniques have been added to its usual pharmacological and physiotherapeutic treatment. Despite the abundant evidence that addresses psychosocial factors as clear mediators in the perception of pain, the use of psychological techniques for pain management in competitive athletes, and more especially in competitive athletes with physical disabilities, is scarce. The purpose of this study was to ascertain the perception of high-level competitive athletes with physical disability and sports agents (coaches, physiotherapists and psychologists).

DETAILED DESCRIPTION:
Qualitative study with in-depth interviews to find out the perception of sports agents (coaches, physiotherapists and psychologists) and athletes on how pain can affect the development of the sports career and to determine what techniques are known and/or implemented by sports agents (coaches, physiotherapists and psychologists) and athletes to manage pain.

ELIGIBILITY:
Inclusion Criteria:

For the athlete:

* Physical disability.
* Participate in high performance competition
* Aged between 15 and 55 years old;

For the sports agents:

* To exercise their profession with high performance athletes with physical disabilities

Exclusion Criteria:

* Not meeting the above requirements

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A total of 20 participants were interviewed on a voluntary basis (7 competitive athletes with physical disabilities, 4 physiotherapists, 5 coaches and 4 psychologists) after being informed of the research objectives. The sports agents (coaches, physiotherapists and psychologists) were active and worked with high-level athletes in their professional field. As for the athletes, all were active except one, who had been retired for eight years, and took part in national and international competitions and Paralympic Games in their respective sports disciplines. All of them belonged to the Spanish Sports Federation for People with Physical Disabilities (FEDDF)
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-01-16 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
Perception of pain in competitive athletes with physical disabilities and techniques for its management.(Qualitative methodology). | 2 months
  This research focuses on the subjective reality of individuals regarding their life experiences of how pain can affect a sporting career. It was based on a relativistic ontology, situated in an overlapping phenomenological and interpretative epistemology.The organisation of the information collected was carried out with "Nuevo NVivo" text processing software. The codes extracted from the thematic analysis were entered. Followed by a thematic analysis of their content and according to the specific objectives of the study. The steps followed were those proposed by Braun and Clarke (2006). Two types of triangulation were applied (Flick, 2014): investigator and data triangulation.
  Pain has a negative impact on the athlete's sporting career: directly or indirectly through the psychological consequences. Athletes perceive that support of a psychologist are performance oriented and not pain management.

CONTACTS AND LOCATIONS:
Overall Officials: María I. Barriopedro, PhD in Psychology, Study Director — Universidad Politecnica de Madrid
Locations (1):
- Universidad Politécnica de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No